CLINICAL TRIAL: NCT06491589
Title: Feasibility and Outcomes of Endovascular Aneurysm Repairs (EVARs) Without Arterial Line Monitoring
Status: Not yet recruiting | Type: Observational
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Loukman Ghouti, Principal investigator, Nova Scotia Health Authority
Other Study IDs: 1030377
Record Dates: First submitted 2024-06-20; First posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: abdominal aortic aneurysm; EVAR; Arterial monitoring
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: EVAR with arterial line monitoring
- Group B: EVAR with no arterial line monitoring

SUMMARY:
Endovascular Aortic Aneurysm Repairs (EVARs) are typically performed with arterial line monitoring, however our institution has successfully omitted this practice in select cases without complications or patient safety concerns. To investigate this further, our planned study will compare patients undergoing EVAR with and without arterial line monitoring. Data will be collected on pre-operative characteristics (patient age, sex, comorbidities), intraoperative details (procedural time, need for emergent intra-operative arterial monitoring or blood draws), and postoperative outcomes (complications, time in post-operative recovery unit). Operating room staff satisfaction and acceptability will be measured using a survey developed by our team. The findings from this study hold promise for improvement the treatment of aortic aneurysms, as well as enhancing patient safety and experience.

DETAILED DESCRIPTION:
The management of aortic aneurysms has undergone a remarkable transformation in recent years, moving from traditional open surgical approaches to minimally invasive endovascular techniques. Historically, aortic aneurysm repair was primarily conducted through open aneurysm repair (OAR), involving a large abdominal incision to access the diseased segment of the aorta directly. Although effective, OAR was characterized by extensive surgical trauma, prolonged operative times, and significant physiological disturbances, often requiring intensive care stays with associated morbidity and mortality. In recent decades, the landscape has greatly shifted such that aortic aneurysm repair has now become a streamlined procedure, with some medical centers offering endovascular repair as day procedures, and allowing most patients to return home the following day.

Endovascular Aneurysm Repair (EVAR) has been pivotal in this transformation, providing minimally invasive alternatives to traditional open surgery. Unlike conventional approaches, EVAR involves repairing aneurysms without a large laparotomy incision and aortic clamping, using instead stent grafts delivered from within the vessel to reinforce weakened sections of the aorta. This method offers numerous advantages over conventional surgery, including reduced surgical trauma and shorter recovery times. Historically, EVARs required general anesthesia and bilateral femoral surgical exposure. However, recent innovations, such as percutaneously inserted lower-profile devices and the use of local anesthesia, have further simplified the procedure, mitigating the complexities associated with general anesthesia induction and maintenance.

Usually, following the patient's entry into the operating room for an EVAR procedure, they are provided with an arterial line. Arterial lines ('art' lines) allow continuous monitoring of blood pressure, providing beat-to-beat measurements. They also offer a convenient method for obtaining arterial blood samples, eliminating the need for multiple needle punctures. Despite their utility, arterial lines carry potential complications (incidence rate of 1% for both minor and major complications across radial, femoral, and axillary artery cannulations among adult patients), including infection, thrombosis, vasospasm, hematoma formation, and air embolism. Inserting an arterial line also extends the procedure time, contingent on factors such as patient anatomy and physician expertise. Patient perception of arterial lines may vary, with some finding the insertion uncomfortable, particularly during initial placement and securing.

At our institution, standard EVARs are preferentially performed with a "simplest practice possible" approach. This idea removes any unnecessary instrumentation of the patient, while still prioritizing patient safety. Our approach so far includes omitting urinary catheterization, employing a percutaneous approach and performing the surgery under local anesthesia. In an effort to advance our understanding and optimize patient care, our institution has explored the possibility of EVARs without arterial line monitoring. Through collaborative discussions involving surgical, anesthesia, and nursing teams, patients deemed candidates have undergone EVAR procedures without arterial monitoring. In cases where beat-to-beat monitoring was necessary intra-operatively, a transducer connected to the femoral arterial sheath was used to provide information equivalent to traditional arterial lines. Similarly, if an arterial blood sample was required, it was obtained directly from the arterial sheath.

This novel approach, though not yet described in literature, holds promise for improving procedural efficiency and patient outcomes. Omitting arterial lines could potentially streamline procedures, enhance patient satisfaction, and reduce complication risks associated with arterial access. Reforming standard-of-care paradigms, whether in clinic or operating room, is a well-established practice in medicine. A similarly innovative approach was undertaken by the Vancouver Heart Team for transcatheter aortic valve replacement (TAVR) procedures. They developed a standardized clinical pathway for safe early discharge after TAVR. Following implementation, retrospective analysis revealed that patients discharged early exhibited more favorable clinical indicators compared to those with standard discharge protocols. This study, one among many, illustrates how simplifying procedures and care standards, while maintaining patient safety, can achieve positive outcomes.

However, several critical questions remain unanswered, including the impact on operating time, complication rates, and acceptance by the treating teams. As such, this proposal seeks to address these uncertainties by investigating the feasibility and outcomes of EVARs without arterial line monitoring. By systematically evaluating this approach, we aim to optimize patient care pathways and enhance procedural efficiency.

ELIGIBILITY:
Inclusion Criteria:

Adult patients undergoing percutaneous EVAR at the Queen Elizabeth II Health Sciences center from June 1st 2024 - May 31st 2025.

Exclusion Criteria:

* Patients requiring surgical femoral exposure.
* Patients requiring fenestrated endografts: these are more complex cases, take a longer duration, usually require a general anesthetic and are at higher risk of arterial rupture, and thus cannot safely be performed without an arterial line.
* Patients undergoing EVAR with an Endologix endograft: there is a small risk of anaphylaxis with the polymer used with the Endologix endograft, and thus the arterial line is required for beat-to-beat monitoring during graft deployment.
* Patients with heavily calcified iliac or femoral arteries: this increases the risk of arterial rupture, and thus requires beat-to-beat arterial monitoring.
* Absence of significant co-morbidities: no severe aortic stenosis (AS) (suspected AS and echo diagnostic criteria: max jet velocity >4.0 m/s, mean gradient >40 mmHg, valve area <1 cm²); No congestive heart failure (CHF) (CHF diagnostic criteria: ejection fraction (EF) below 50% and natriuretic (NT) pro-Brain Natriuretic Peptide (BNP) levels based on the following age-adjusted cutoff limits.

  * Age < 50 years: NT pro-BNP greater than 450 ng/L.
  * Age 50-75 years: NT pro-BNP greater than 900 ng/L.
  * Age > 75 years: NT pro-BNP greater than 1800 ng/L.); Blood pressure below 180/120 on the morning of the operation day; Surgeon and/or anesthesiologist discretion.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients undergoing percutaneous EVAR at the QEII Health Sciences center.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Assess acceptability of no art-line EVAR. | 12 months
  Acceptability (user satisfaction, perceived appropriateness, perceived positive or negative effects on organization) will be determined by a Likert scale survey circulated to treating staff.
Assess technical feasibility of no art-line EVAR. | 12 months
  Technical feasibility (time required for pre-op prep and setup; duration of procedure)
Asess safety of no art-line EVAR. | 12 months
  Although this has already been established to be a safe and viable surgical technique, it would still be interesting to collect data on the incidence of intra-op and post-op complications.

SECONDARY OUTCOMES:
Assess complication rates of no art-line EVAR as compared to traditional EVAR procedures using arterial line monitoring. | 12 months
  Assess the overall complication rates (incidence) of the no art-line approach to EVAR.

CONTACTS AND LOCATIONS:
Overall Officials: Loukman Ghouti, Principal Investigator — Dalhousie University
Locations (1):
- QEII Health Sciences Center, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: Undecided
This discussion has not been broached yet.

REFERENCES:
- [Background] Dunn K, Jessula S, Herman CR, Smith M, Lee MS, Casey P. Safety and effectiveness of single ProGlide vascular access in patients undergoing endovascular aneurysm repair. J Vasc Surg. 2020 Dec;72(6):1946-1951. doi: 10.1016/j.jvs.2020.03.028. Epub 2020 Apr 8. PMID 32276013
- [Background] Jessula S, Cote C, Khoury M, DeCarlo C, Bellomo TR, Grant-Gorveatt A, Herman C, Smith M, Dua A, Eagleton M, Casey P, Zacharias N. Local Anesthesia for Endovascular Repair of Abdominal Aortic Aneurysm Allows for Accurate Graft Deployment with Durable Results. Ann Vasc Surg. 2024 May;102:64-73. doi: 10.1016/j.avsg.2023.11.033. Epub 2024 Jan 30. PMID 38301848